CLINICAL TRIAL: NCT02070133
Title: Pilot Study on the Efficacy of Statins for the Treatment of Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy of Simvastatin for the Treatment of COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Son Dureta (Other)
Collaborators: Fundació d'investigació Sanitària de les Illes Balears (Other Government); Cimera (Network)
Responsible Party: Principal Investigator, Ernest Sala, Medical Doctor, Hospital Son Espases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC08/00123
Record Dates: First submitted 2013-10-14; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Bronchitis; Statins; Endothelial dysfunction; Systemic inflammation; BODE index; Uric acid; Vascular growth factors
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Experimental): Patients with COPD will receive simvastatin 40 mg once a day for 12 weeks
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Patients with COPD will receive placebo once a day during 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40 mg once a day during 12 weeks
  Arms: Simvastatin
Drug: Placebo — Placebo once a day during 12 weeks
  Arms: Placebo

SUMMARY:
To evaluate in patients with stable Chronic Obstructive Pulmonary Disease (COPD) the efficacy of statins (simvastatin) on: (1) endothelial function; (2) systemic inflammation; (3)BODE (B: body mass , O: bronchial obstruction, D: dyspnea and, E: exercise tolerance) index; (4) Uric acid; and, (5)vascular growth factors. Design: a 12 weeks randomized (1:1), double-blind, placebo control study. Population: 18 males with stable COPD between 40-80 years of age, exsmokers, with Forced expiratory volume in one second (FEV1) between 30 and 80% predicted post-bronchodilation.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD between 40-80 years of age, exsmokers, with FEV1 lower that 80% predicted post-bronchodilation.

Exclusion Criteria:

* Severe co-morbidity (advanced-stage cancer, tuberculosis affecting more than a third of the total lung parenchyma, pneumonectomy, pneumoconiosis, left cardiac failure previously reported, known cardiopathy with ventricular dysfunction (ejection fraction < 45%) or any cardiovascular disease, Diabetes Mellitus treated with insulin, Hypercholesterolemia, Chronic inflammatory diseases (asthma, rheumatoid arthritis, lung fibrosis, autoimmune diseases), Treatment with systemic steroid, non steroidal anti-inflammatory drugs or stains within 3 months prior to inclusion.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-05; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Endothelial Dysfunction (Arterial Stiffness) | Day 1 and day 84 (end of of week 12)

SECONDARY OUTCOMES:
Systemic inflammation | Day 1 and day 84 (end of of week 12)
BODE index | Day 1 and day 84 (end of of week 12)
Uric acid | Day 1 and day 84 (end of of week 12)
Vascular growth factors | Day 1 and day 84 (end of of week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Sala, MD, Principal Investigator — Hospital Son Espases, Palma Mallorca
Locations (2):
- Spain (2):
  - Fundacio Caubet-CIMERA, Bunyola, Balearic Islands
  - Hospital Son Espases, Palma Mallorca, Balearic Islands